CLINICAL TRIAL: NCT01537640
Title: A Randomized, Double-Blind, Parallel Group Study of the Pharmacokinetics, Safety, and Tolerability of Two Different SAR231893 Drug Products After Administration of a Single Subcutaneous Dose to Healthy Subjects
Brief Title: Comparison of the Pharmacokinetics and Safety of Two SAR231893 (REGN668) Drug Products in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PKM12350; U1111-1119-3152 (Other: UTN)
Record Dates: First submitted 2012-02-17; First posted 2012-02-23 (Estimated); Last update posted 2013-12-06 (Estimated); Status verified 2012-07

CONDITIONS: Healthy
MeSH Terms: interventions — dupilumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- SAR231893 (REGN668) Drug Product (DP) 1 (Experimental): SAR231893 (REGN668) Drug Product 1 in a single subcutaneous injection
  Interventions: Biological: SAR231893 (REGN668) DP1
- SAR231893 (REGN668) Drug Product (DP) 2 (Experimental): SAR231893 (REGN668) Drug Product 2 in a single subcutaneous injection
  Interventions: Biological: SAR231893 (REGN668) DP2

INTERVENTIONS:
Biological: SAR231893 (REGN668) DP1 — Pharmaceutical form:solution Route of administration: subcutaneous
  Arms: SAR231893 (REGN668) Drug Product (DP) 1
Biological: SAR231893 (REGN668) DP2 — Pharmaceutical form:solution Route of administration: subcutaneous
  Arms: SAR231893 (REGN668) Drug Product (DP) 2

SUMMARY:
Primary Objective:

To determine and compare the pharmacokinetic (PK) profiles of 2 different SAR231893 (REGN668) drug products after administration of a single subcutaneous (SC) dose

Secondary Objective:

To determine and compare the safety and tolerability of the 2 SAR231893 (REGN668) drug products after administration of a single SC dose

DETAILED DESCRIPTION:
The duration of the study for each subject is 8-11 weeks broken down as follows:

* Screening: 2 to 21 days,
* Treatment: 1 day (2 overnight stays at the study site),
* Follow-up: up to 2 months after dosing.

ELIGIBILITY:
Inclusion criteria:

* Healthy male and female subjects between 18 and 45 years of age

Exclusion criteria:

* Presence or history of drug hypersensitivity or allergic disease
* History or presence of dermatological disorders
* Fever or persistent chronic or active recurring infection requiring treatment within 4 weeks prior to screening, or history of frequent recurrent infections
* Prior opportunistic infections within 6 months before inclusion
* History or presence of listeriosis or tuberculosis
* Any vaccination within 3 months (1 month for influenza vaccine) before inclusion
* Any biologics given within 4 months before inclusion
* Recent history of a parasitic infection or travel to a parasitic endemic area within 6 months prior to screening

The above information is not intended to contain all considerations relevant to a subject's potential participation in a clinical trial.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2012-02; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Assessment of serum concentrations of SAR231893 (REGN668) | Up to 57 Days

SECONDARY OUTCOMES:
Pain evaluation at injection site using Visual Analog Scale (VAS) | Up to 8 Days
Erythema at injection site by measuring diameter | Up to 8 Days
Edema at injection site by measuring diameter | Up to 8 Days
Number of participants experiencing adverse events | Up to 57 Days

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Investigational Site Number 840001, Daytona Beach, Florida, United States

REFERENCES:
- [Derived] Li Z, Radin A, Li M, Hamilton JD, Kajiwara M, Davis JD, Takahashi Y, Hasegawa S, Ming JE, DiCioccio AT, Li Y, Kovalenko P, Lu Q, Ortemann-Renon C, Ardeleanu M, Swanson BN. Pharmacokinetics, Pharmacodynamics, Safety, and Tolerability of Dupilumab in Healthy Adult Subjects. Clin Pharmacol Drug Dev. 2020 Aug;9(6):742-755. doi: 10.1002/cpdd.798. Epub 2020 Apr 29. PMID 32348036